CLINICAL TRIAL: NCT02432027
Title: A Single-Center, Randomized, Observer Blind, Vehicle- and Comparator-controlled Trial to Evaluate the Antipsoriatic Efficacy and Safety of Topical Formulations of C-82 in a Psoriasis Plaque Test
Brief Title: Trial to Evaluate Topical C-82 in a Psoriasis Plaque Test
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prism Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRI-C-82T-2101
Record Dates: First submitted 2015-04-28; First posted 2015-05-01 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2015-10

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- IMP 1 (Experimental): C-82 Topical Gel, 1%
  Interventions: Drug: C-82 Topical Gel, 1%
- IMP 2 (Placebo Comparator): C-82 Topical Gel, placebo
  Interventions: Drug: C-82 Topical Gel, Placebo
- IMP 3 (Active Comparator): Daivonex cream
  Interventions: Drug: Daivonex cream
- IMP 4 (Active Comparator): Diprosis gel
  Interventions: Drug: Diprosis gel

INTERVENTIONS:
Drug: C-82 Topical Gel, Placebo — placebo
  Arms: IMP 2
Drug: C-82 Topical Gel, 1% — active
  Arms: IMP 1
Drug: Daivonex cream — comparator
  Other Names: calcipotriol 50mcg/g
  Arms: IMP 3
Drug: Diprosis gel — comparator
  Other Names: betamethasone, 0.5 mg/g
  Arms: IMP 4

SUMMARY:
Evaluate the effects of topical C-82 in a psoriasis plaque test.

DETAILED DESCRIPTION:
The primary objective of this trial is to evaluate antipsoriatic efficacy of the C-82 topical gel compared with vehicle by measurement of the thickness of the Echo Lucent Band (ELB) of the psoriatic infiltrate using 20 MHz sonography. To gain additional information about possible efficacy the change of the test fields compared to untreated plaque will be clinically assessed by visual scoring.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate chronic stable plaque type psoriasis
* plaques thickness of at least 200 µm
* lesion(s) on the trunk or extremities (excluding palms/soles)
* skin must be without disease findings

Exclusion Criteria:

* other skin disease
* psoriasis guttata, psoriasis punctata, psoriasis erythrodermatica, psoriasis arthropathica and pustular psoriasis
* treatment with any locally acting medications (including anti-psoriatics like vitamin D analogues, dithranol) within 2 weeks preceding and during the trial
* treatment with any systemic medications (including anti-psoriatics like corticosteroids, cytostatics or retinoids) or medications which are known to provoke or aggravate psoriasis (e.g. beta-blocker, anti-malarial drugs, lithium) or phototherapy/PUVA within 4 weeks preceding and during the trial
* treatment with any biologics within 3 months preceding and during the trial
* known allergic reactions, irritations or sensitivity to the active ingredients or other components of the investigational products (e.g. Carbomere 940, propylene glycol)
* drug or alcohol abuse
* symptoms of a clinically significant illness within 4 preceding and during the trial
* participation another clinical trial within 4 weeks of this clinical trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
antipsoriatic efficacy of the C-82 topical gel compared with vehicle by measurement of the thickness of the Echo Lucent Band (ELB) of the psoriatic infiltrate | day 12

SECONDARY OUTCOMES:
antipsoriatic efficacy compared to control by clinical assessment using a 5-point score. | Day 8 & Day 12
number of subjects with adverse events | daily through Day 12

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Theis, MD, Principal Investigator — Klinische Forschung Schwerin GmbH
Locations (1):
- Schwerin, Germany